CLINICAL TRIAL: NCT01407315
Title: Accuracy, Reliability and Safety of GlucoMen®Day, a New Generation Microdialysis Continuous Glucose Monitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Menarini Group (Industry)
Responsible Party: Principal Investigator, Pieber Thomas, MD, MD, Prof. of Medicine, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GMD_03
Record Dates: First submitted 2011-05-23; First posted 2011-08-02 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Type 1 Diabetes
Keywords: Continuous subcutaneous glucose monitoring; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GlucoMenDay - Multiple sampling (A) (Experimental)
  Interventions: Device: GlucoMenDay
- GlucoMenDay - Meal/Insulin test (B) (Experimental)
  Interventions: Device: GlucoMenDay

INTERVENTIONS:
Device: GlucoMenDay — Subjects will receive a standardized lunch (100 g of CHO), administration of insulin will be performed by the subject based on insulin to carbohydrate ratio.
  An intravenous catheter will be inserted in one forearm and venous sampling will start 1 hour after lunch ingestion. Arterialized-venous blood sampling will be performed every 15 minutes for a period of two hours. Samples will be analyzed for glucose using the Super GL; concomitantly capillary measurements using the GlucoCard G Meter will be performed.
  This procedure can be performed on days 3-4 of monitoring; each subject randomized to Procedure A undergoes this procedure once.
  Other Names: Continuous Glucose Monitoring
  Arms: GlucoMenDay - Multiple sampling (A)
Device: GlucoMenDay — Subjects will receive a standard breakfast (75g CHO), the usual morning insulin dose will be post-poned. An increased dose of rapid-acting insulin analogue aiming to produce minor hypoglycaemia based on insulin to carbohydrate ratio will be injected subcutaneously. Arterialized-venous sampling will be performed every 10 minutes for a period of two hours.
  Samples will be analyzed for glucose using the Super GL; concomitantly, capillary measurements using the GlucoCard G Meter will be performed.
  This procedure will be performed on days 2 and 4 of monitoring; each subject randomized to Procedure B undergoes this procedure twice.
  Other Names: Continuous Glucose Monitoring
  Arms: GlucoMenDay - Meal/Insulin test (B)

SUMMARY:
Monocenter single-arm, prospective clinical study in 20 type 1 diabetic subjects, equipped with the GlucoMen®Day system, over up to 100 hours observation after implantation of the microdialysis probe. Different meal/hypo procedures will be performed at the study centre.

DETAILED DESCRIPTION:
This is a monocenter single-arm, prospective clinical study in 20 type 1 diabetic subjects, who will be equipped with the GlucoMen®Day system.

Each subject will be investigated for up to 100 hours after implantation of the microdialysis probe.

In order to verify the clinical effectiveness of the GlucoMenDay the subjects will be asked to perform a total of six self testing measurements per day using the GlucoCard G-Meter according to the following scheme:

* before breakfast
* before lunch
* 60-120 minutes after lunch
* before dinner
* 60-120 minutes after dinner
* at 3 AM

Subjects will be asked to come to the research facility every day to obtain a venous blood sample and to check system functioning.

Subjects will be randomized either to Procedure A - Multiple sampling or Procedure B - Meal/Insulin test.

Procedure A - Multiple sampling:

This procedure can be performed at days 2-4 of the study period. Subjects will receive a standardized lunch (100 g of CHO), administration of insulin will be performed by the subject based on insulin to carbohydrate ratio. An intravenous catheter will be inserted in one forearm and venous sampling will start 1 hour after lunch ingestion. Arterialized-venous blood sampling will be performed every 15 minutes for a period of two hours. Samples will be analyzed for glucose using the Super GL; concomitantly capillary measurements using the GlucoCard G Meter will be performed.

Procedure B - Meal/Insulin test:

This procedure will be performed on days 2 and four of the experiment. Subjects randomized to procedure B will be asked to undergo this investigation twice.

Subjects will receive a standard breakfast (75g CHO), the usual morning insulin dose will be post-poned. An increased dose of rapid-acting insulin analogue aiming to produce minor hypoglycaemia based on insulin to carbohydrate ratio will be injected subcutaneously. Arterialized-venous sampling will be performed every 10 minutes for a period of two hours.

Samples will be analyzed for glucose using the Super GL; concomitantly, capillary measurements using the GlucoCard G Meter will be performed.

On day 5 subjects will return to the clinical trial unit for collection of a final blood sample and removal of the device.

Subjects will be asked to come to the research facility at 48 and 72 hours after removal of the device for an evaluation of local site reactions.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of type-1-diabetes
* Ability to provide informed consent
* Age 18-75 years

Exclusion Criteria:

* Subjects under anti-coagulant treatments
* Alcoholism
* Body mass index (BMI) > 32 kg/m2
* Inability to adhere to the protocol or to attend the required follow- up visits and tests
* Diseases or conditions of the abdominal wall which, in the opinion of Clinician might contraindicate the insertion of the hypodermic needle into the subcutaneous tissue
* Legal incapacity and/or other circumstances rendering the subject unable to understand the nature, scope and possible consequences of the study
* Any serious medical conditions or disability, which in the opinion of the investigator, would interfere with treatment or assessment or preclude completion of the study
* Subjects currently participating in a clinical study
* Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of the GlucoMenDay | 1 week
  Assessed by methods such as the Clarke Error Grid Analysis (EGA), CG-EGA, MARD, MAD

SECONDARY OUTCOMES:
Safety of the GlucoMenDay System | 1 week
  Assessment of patients with local skin reaction at insertion site after 100 hours of continuous monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria